CLINICAL TRIAL: NCT01622582
Title: Engraftment Syndrome After Autologous Stem Cell Transplant: Retrospective Review in Patients With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: UARK 2008-30
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma, Engraftment syndrome
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Engraftment Syndrome after Autologous Stem Cell Transplant: Retrospective Review in Patients with Multiple Myeloma

DETAILED DESCRIPTION:
A retrospective chart review series will be performed fpr subjects enrolled from 1/1/2006.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple Myeloma, developing engraftment syndrome

Exclusion Criteria:

* Patients with Multiple Myeloma, with no features of engraftment syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma, developing engraftment syndrome
Sampling Method: Non-Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2006-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
number of patients developing Engraftment syndrome following stem cell transplant | 6 months post-transplant
  A retrospective review where subjects medical records are studied for development of engraftment syndrome 6 months after stem cell transplant

CONTACTS AND LOCATIONS:
Overall Officials: Senu Apewokin, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States